CLINICAL TRIAL: NCT04344314
Title: A Randomized Controlled Post-market Study to Assess the Impact of Peripheral Intravenous Catheter Length and Gauge on Catheter Indwell Duration and Haemolysis in Human Participants Using a Bilateral, Cephalic Vein Cannulation Model
Brief Title: Impact of PIVC Length and Gauge on Catheter Indwell Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Becton, Dickinson and Company (Industry)
Collaborators: Griffith University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: BDT-PIVCAU001
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-07

CONDITIONS: Indication for Peripheral Intravenous Catheterisation

STUDY DESIGN:
Intervention Model Description: Randomised, controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Small gauge arm (Other): 2 PIVCs of same gauge (22G) and different lengths
  Interventions: Device: Peripheral Intravenous Catheter
- Large gauge arm (Other): 2 PIVCs of same gauge (20G) and different lengths
  Interventions: Device: Peripheral Intravenous Catheter

INTERVENTIONS:
Device: Peripheral Intravenous Catheter — Randomised controlled

SUMMARY:
This is a single-centre, open-label, multi-visit study design, in 40 healthy participants, randomized by gauge of peripheral intravenous catheter (PIVC) device into the lower arm cephalic vein of both arms.

The purpose of this study is to assess impact of catheter length and gauge on PIVC indwell time over a 72 hour period. This study will also evaluate the incidence of haemolysis using blood draws from the PIVC.

DETAILED DESCRIPTION:
The study aims to provide preliminary information on the performance of the peripheral intravenous catheter (PIVC) device,

* assess how blood collection through different catheters over time effects device performance, and
* assess the quality of the blood that is collected through those catheters. Four variations of the Becton Dickinson (BD) Nexiva PIVC will be used in this study. Participants will be randomised by gauge of peripheral intravenous catheter (PIVC) device into the lower arm cephalic vein of both arms. PIVC indwell time will be monitored up to 72 hrs (removal at 72 hrs or upon inability to flush/aspirate). Blood will be collected Day 1 throughout the remainder of indwell time.

Each participant will complete 6 visits: a Screening Visit (V1), PIVC in situ (V2-V5) and follow-up (V6).

The in-situ catheter positions will be compared to the expected tip position based on the catheter lengths. Blood collected will be analysed for haemolysis.

As both device length and gauge are expected to influence haemolysis the study design enables evaluation of both design features.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* 18-65 years of age
* Not pregnant at time of recruitment within 48 hrs Day 1 procedures (self-reported)
* Normal coagulation results (prothrombin time 13-17 sec; activated partial thromboplastin time 27-37 sec)
* Normal platelet aggregation results for Adenosine DiPhosphate (ADP), Thrombin Receptor Activating Peptide (TRAP), and collagen induced maximal amplitude (>70% amplitude over 6 mins)
* Target cephalic veins readily cannulatable (i.e., ≥ ~2.55 mm to obtain C/V ratio less than 45% as indicated by standard 52 of the Intraevenous Nursing Standards (INS) guidelines
* Able and willing to provide verbal and written consent
* Must be an Australian citizen with current Medicare card

Exclusion Criteria:

* History of pro coagulative state/condition (e.g. previous deep vein thrombosis
* Current hypertension (e.g., systolic >139 OR diastolic >89 mmHg)
* Currently on any anti-coagulant or platelet inhibitor medication. Use of NSAIDs and aspirin will be documented however not exclusionary.
* Hemophilia or any current or history of bleeding disorder or tendency
* Presence or report of current blood borne disease/infection (e.g. hepatitis, HIV, leukemia, lymphoma)
* Difficult vascular access (i.e., vein must be readily palpable and cannulatable - no less than ~2.55 mm diameter to maintain ≤45% C/V ratio) as indicated by standard 52 of the INS guidelines
* Allergy or sensitivity to chlorhexidine gluconate, isopropyl alcohol, latex, or skin adhesives
* BMI <18.5 kg/m2 or ≥35 kg/m2
* Positive results for the urine drug screen at screening or check-in (including opiates, methadone, cocaine, amphetamines)
* History or presence of alcoholism (self-reported) or drug abuse within the past 2 years
* A current or previous medical, physical, mental/cognitive disorders or anatomical conditions that, in the opinion of the investigator, would place the patient at risk, would make them unable to perform study procedures or has the potential to confound interpretation of the study results. (e.g., musculo-skeletal injury, chronic back pain)
* Employed by Becton Dickinson, Teleflex Medical, Smiths Medical or B Braun (conflict of interest)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-08-31 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Griffith University, Gold Coast, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 enrolled and randomized subjects
Units Other Than Participants: arms
Groups:
- PIVC 22G, 1 Inch Length: One participant receives 2 Peripheral Intravenous Catheters (PIVC) with the same Gauge (22G), one in each arm.
  The length of the catheter is different in each arm, in this case: 1 Inch.
  Choice of catheter size and length is randomized per participant, as well as which arm is first catharized.
- PIVC 22G, 1.75 Inch Length: One participant receives 2 Peripheral Intravenous Catheters (PIVC) with the same Gauge (22G), one in each arm.
  The length of the catheter is different in each arm, in this case: 1.75 Inch.
  Choice of catheter size and length is randomized per participant, as well as which arm is first catharized.
- PIVC 20G, 1 Inch Length: One participant receives 2 Peripheral Intravenous Catheters (PIVC) with the same Gauge (20G), one in each arm.
  The length of the catheter is different in each arm, in this case: 1 Inch.
  Choice of catheter size and length is randomized per participant, as well as which arm is first catharized.
- PIVC 20G, 1.75 Inch Length: One participant receives 2 Peripheral Intravenous Catheters (PIVC) with the same Gauge (20G), one in each arm.
  The length of the catheter is different in each arm, in this case: 1.75 Inch.
  Choice of catheter size and length is randomized per participant, as well as which arm is first catharized.
Period: Overall Study
Arm/Group | PIVC 22G, 1 Inch Length | PIVC 22G, 1.75 Inch Length | PIVC 20G, 1 Inch Length | PIVC 20G, 1.75 Inch Length
Started | 19; 19 arms | 19; 19 arms | 21; 21 arms | 21; 21 arms
Completed | 19; 19 arms | 19; 19 arms | 21; 21 arms | 21; 21 arms
Not Completed | 0; 0 arms | 0; 0 arms | 0; 0 arms | 0; 0 arms

BASELINE CHARACTERISTICS:
Groups:
- Small Gauge: 2 PIVCs of same gauge (22G) and different lengths
  Peripheral Intravenous Catheter: Randomised controlled
- Large Gauge: 2 PIVCs of same gauge (20G) and different lengths
  Peripheral Intravenous Catheter: Randomised controlled
- Total: Total of all reporting groups
Arm/Group | Small Gauge | Large Gauge | Total
Number analyzed (Participants) | 19 | 21 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.58 (8.82) | 32.76 (13.12) | 30.3 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 6 | 7 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11 | 12 | 23
  Unknown | 0 | 5 | 5
  Asian | 4 | 0 | 4
  Asian, White | 2 | 0 | 2
  Native Hawaiian or other Pacific Islander | 0 | 2 | 2
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 19 | 21 | 40
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.09 (3.65) | 26.84 (5.22) | 26.01 (4.57)
Recent use of analgesics [Count of Participants; unit: Participants]
  Recent use of analgetic | 6 | 2 | 8
  No recent use of analgetic | 13 | 19 | 32
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 115.83 (10.75) | 117.90 (10.02) | 116.92 (10.29)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 76.42 (8.09) | 76.71 (7.40) | 76.58 (7.46)
O2 saturation [Mean (Standard Deviation); unit: Percentage of oxygen in blood] | 97.89 (1.05) | 97.71 (1.23) | 97.80 (1.14)

OUTCOME MEASURES:

1. Primary Outcome: Patent Indwell Time Between PIVCs of Different Length and Gauge.
Description: Catheter indwell time for each PIVC, expressed in hours
Time Frame: 72 hrs
Population: After screening and enrollment, participants will be randomized in order of their enrollment to either 20 or 22G of the BD NexivaTM PIVC and order of placement location (left or right arm first). The participant will have both the 1 inch and 1.75 inch PIVCs inserted on Study Day 1 (Visit 2), one into each arm. After successful insertion into the lower cephalic vein of the selected arm, the site will be regularly accessed (twice daily) for phlebotomy and then flushed.
Measure: Mean (Standard Deviation); unit: hours
Groups:
- PIVC 22G, 1 Inch Length: small gauge, shorter catheter
- PIVC 22G, 1.75 Inch Length: small gauge, longer catheter
- PIVC 20G, 1 Inch Length: large gauge, smaller catheter
- PIVC 20G, 1.75 Inch Length: large gauge, larger catheter
Arm/Group | PIVC 22G, 1 Inch Length | PIVC 22G, 1.75 Inch Length | PIVC 20G, 1 Inch Length | PIVC 20G, 1.75 Inch Length
Number analyzed (Participants) | 19 | 19 | 21 | 21
hours | 40.19 (25.34) | 42.96 (22.04) | 35.91 (25.55) | 36.91 (21.36)

2. Secondary Outcome: Number of Participants With Haemolysis Occurrence Based on Blood Collection Device and Catheter Device Configuration
Description: Haemolysis: Frequency of occurrence
Time Frame: 72 hrs
Measure: Count of Units; unit: arms
Units Other Than Participants: arms
Arm/Group | PIVC 22G, 1 Inch Length | PIVC 22G, 1.75 Inch Length | PIVC 20G, 1 Inch Length | PIVC 20G, 1.75 Inch Length
Number analyzed (Participants) | 19 | 19 | 21 | 21
Number analyzed (arms) | 19 | 19 | 21 | 21
arms
  Visual haemolysis, 2 mL collection tube | 0 | 0 | 0 | 0
  Visual haemolysis, 6 mL collection tube | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse Events are collected from time of enrollment until catheter removal (max 72 hours indwell time)
Description: Adverse Events are systematically collected during the study visits and a Clinical Research Associate actively reviewed the patient medical records for any occurred events.
Groups:
- PIVC 22G, 1 Inch Length: Adverse Events are presented for all participants within the group of participants receiving the small gauge catheter of 22G, for 1 Inch catheter length.
- PIVC 22G, 1.75 Inch Length: Adverse Events are presented for all participants within the group of participants receiving the large gauge catheter of 22G, for 1.75 Inch catheter length.
- PIVC 20G, 1 Inch Length: Adverse Events are presented for all participants within the group of participants receiving the large gauge catheter of 20G, for 1 Inch catheter length.
- PIVC 20G, 1.75 Inch Length: Adverse Events are presented for all participants within the group of participants receiving the large gauge catheter of 20G, for 1.75 Inch catheter length.
Arm/Group | PIVC 22G, 1 Inch Length | PIVC 22G, 1.75 Inch Length | PIVC 20G, 1 Inch Length | PIVC 20G, 1.75 Inch Length
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21 | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 1/19 | 1/19 | 11/21 | 8/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PIVC 22G, 1 Inch Length (N=19) | PIVC 22G, 1.75 Inch Length (N=19) | PIVC 20G, 1 Inch Length (N=21) | PIVC 20G, 1.75 Inch Length (N=21)
Thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Inflammatory pain (General disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
Venous thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — This AE cannot be attributed to either catheter length - the only thing that is certain is that it happened in the 20G group
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This AE cannot be attributed to either catheter length - the only thing that is certain is that it happened in the 20G group
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — This AE cannot be attributed to either catheter length - the only thing that is certain is that it happened in the 20G group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT04344314/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-17): https://cdn.clinicaltrials.gov/large-docs/14/NCT04344314/SAP_001.pdf